CLINICAL TRIAL: NCT01068665
Title: A Trial Comparing Efficacy and Safety of NN1250 and Insulin Glargine in Subjects With Type 2 Diabetes (BEGIN™: LOW VOLUME)
Brief Title: Comparison of NN1250 With Insulin Glargine in Subjects With Type 2 Diabetes
Acronym: BEGIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3672; 2009-010662-28 (EudraCT Number); U1111-1112-8977 (Other: WHO)
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Results first posted 2015-11-13 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg 200 U/mL OD (Experimental)
  Interventions: Drug: insulin degludec
- IGlar OD (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec — Injected subcutaneously (under the skin) once daily. Dose was individually adjusted.
  Arms: IDeg 200 U/mL OD
Drug: insulin glargine — Injected subcutaneously (under the skin) once daily. Dose was individually adjusted.
  Arms: IGlar OD

SUMMARY:
This trial is conducted in South Africa, Europe and North America. The aim of this trial is to compare efficacy and safety of NN1250 (insulin degludec (IDeg)) with insulin glargine (IGlar), as add-on to subject's ongoing treatment with metformin and/or dipeptyl peptidase 4 (DPP-4) inhibitors, in patients with type 2 diabetes being treated with oral anti-diabetic drugs (OADs) qualifying for intensified treatment.

ELIGIBILITY:
Inclusion Criteria:

* Insulin naïve subject (allowed are: previous short term insulin treatment up to 14 days; Treatment during hospitalisation or during gestational diabetes is allowed for periods longer than 14 days)
* Current treatment: metformin monotherapy or metformin in any combination with an insulin secretagogue (sulfonylurea or glinide), DPP-4 inhibitor, alpha-glucosidase-inhibitors (acarbose) with unchanged dosing for at least 3 months prior to visit 1 with the minimum doses stated: -Metformin: alone or in combination (including fixed combination) 1500 mg daily, or maximum tolerated dose (at least 1000 mg daily) -Insulin secretagogue (sulfonylurea or glinide): minimum half of the daily maximal dose according to local labelling -DPP-4 inhibitor: minimum half of the daily maximal dose according to local labelling - alpha-glucosidase-inhibitors (acarbose): minimum half of the daily maximal dose or maximum tolerated dose
* HbA1c 7.0-10.0 % (both inclusive) by central laboratory analysis
* Body Mass Index (BMI) maximum 45.0 kg/m^2
* Type 2 diabetes (diagnosed clinically) for at least 6 months
* Ability and willingness to adhere to the protocol including performance of self monitored plasma glucose (SMPG) profiles according to the protocol

Exclusion Criteria:

* Use within the last 3 months prior to Visit 1 of: thiazoledinediones (TZDs), exenatide or liraglutide
* Cardiovascular disease, within the last 6 months prior to Visit 1, defined as: stroke; decompensated heart failure New York Heart Association (NYHA) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty
* Uncontrolled treated/untreated severe hypertension (systolic blood pressure at least 180 millimetre (mm) mercury (Hg) and/or diastolic blood pressure at least 100 mmHg)
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures according to local requirements [for UK: adequate contraceptive measures are defined as established use of oral, injected or implanted hormonal methods of contraception, sterilisation, intrauterine device or intrauterine system, or consistent use of barrier methods]
* Cancer and medical history of cancer hereof (except basal cell skin cancer or squamous cell skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (109):
- United States (60):
  - Novo Nordisk Investigational Site, Huntsville, Alabama
  - Novo Nordisk Investigational Site, Gilbert, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, Mission Hills, California
  - Novo Nordisk Investigational Site, Montclair, California
  - Novo Nordisk Investigational Site, National City, California
  - Novo Nordisk Investigational Site, Norco, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Valencia, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Longwood, Florida
  - Novo Nordisk Investigational Site, Ocala, Florida
  - Novo Nordisk Investigational Site, Ponte Vedra, Florida
  - Novo Nordisk Investigational Site, Vero Beach, Florida
  - Novo Nordisk Investigational Site, Decatur, Georgia
  - Novo Nordisk Investigational Site, Lawrenceville, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Crystal Lake, Illinois
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Greenfield, Indiana
  - Novo Nordisk Investigational Site, Des Moines, Iowa
  - Novo Nordisk Investigational Site, Madisonville, Kentucky
  - Novo Nordisk Investigational Site, Slidell, Louisiana
  - Novo Nordisk Investigational Site, Greenbelt, Maryland
  - Novo Nordisk Investigational Site, Brockton, Massachusetts
  - Novo Nordisk Investigational Site, Southfield, Michigan
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Biloxi, Mississippi
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Billings, Montana
  - Novo Nordisk Investigational Site, Brick, New Jersey
  - Novo Nordisk Investigational Site, Mine Hill, New Jersey
  - Novo Nordisk Investigational Site, Brooklyn, New York
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Asheboro, North Carolina
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Beaver, Pennsylvania
  - Novo Nordisk Investigational Site, Melrose Park, Pennsylvania
  - Novo Nordisk Investigational Site, Norristown, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Peak, South Carolina
  - Novo Nordisk Investigational Site, DeSoto, Texas
  - Novo Nordisk Investigational Site, El Paso, Texas
  - Novo Nordisk Investigational Site, Killeen, Texas
  - Novo Nordisk Investigational Site, Plano, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, St. George, Utah
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Canada (9):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Langley, British Columbia
  - Novo Nordisk Investigational Site, Cambridge, Ontario
  - Novo Nordisk Investigational Site, Cornwall, Ontario
  - Novo Nordisk Investigational Site, Greater Sudbury, Ontario
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, Mississauga, Ontario
  - Novo Nordisk Investigational Site, Saint Romuald, Quebec
- France (7):
  - Novo Nordisk Investigational Site, Antibes
  - Novo Nordisk Investigational Site, Besançon
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Pointe à Pitre
  - Novo Nordisk Investigational Site, Rennes
  - Novo Nordisk Investigational Site, Sète
  - Novo Nordisk Investigational Site, Vénissieux
- Novo Nordisk Investigational Site, Dublin, Ireland
- Russia (6):
  - Novo Nordisk Investigational Site, Kemerovo
  - Novo Nordisk Investigational Site, Krasnoyarsk
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Voronezh
  - Novo Nordisk Investigational Site, Yekaterinburg
- South Africa (4):
  - Novo Nordisk Investigational Site, East London, Eastern Cape
  - Novo Nordisk Investigational Site, Port Elizabeth, Eastern Cape
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Alberton
- Novo Nordisk Investigational Site, Kiev, Ukraine
- United Kingdom (21):
  - Novo Nordisk Investigational Site, Abergavenny
  - Novo Nordisk Investigational Site, Ashton-under-Lyne
  - Novo Nordisk Investigational Site, Atherstone
  - Novo Nordisk Investigational Site, Ayr
  - Novo Nordisk Investigational Site, Bath
  - Novo Nordisk Investigational Site, Bolton
  - Novo Nordisk Investigational Site, Chester
  - Novo Nordisk Investigational Site, Chorley
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Epworth
  - Novo Nordisk Investigational Site, Harrogate
  - Novo Nordisk Investigational Site, Letchworth Garden City
  - Novo Nordisk Investigational Site, Livingstone
  - Novo Nordisk Investigational Site, Llantrisant
  - Novo Nordisk Investigational Site, Maidstone
  - Novo Nordisk Investigational Site, Oldham
  - Novo Nordisk Investigational Site, Rugby
  - Novo Nordisk Investigational Site, Salford
  - Novo Nordisk Investigational Site, Trowbridge
  - Novo Nordisk Investigational Site, Whitby
  - Novo Nordisk Investigational Site, Wrexham

REFERENCES:
- [Result] Weatherall J, Bloudek L, Buchs S. Budget impact of treating commercially insured type 1 and type 2 diabetes patients in the United States with insulin degludec compared to insulin glargine. Curr Med Res Opin. 2017 Feb;33(2):231-238. doi: 10.1080/03007995.2016.1251893. Epub 2016 Nov 18. PMID 27764979
- [Result] Ratner RE, Gough SC, Mathieu C, Del Prato S, Bode B, Mersebach H, Endahl L, Zinman B. Hypoglycaemia risk with insulin degludec compared with insulin glargine in type 2 and type 1 diabetes: a pre-planned meta-analysis of phase 3 trials. Diabetes Obes Metab. 2013 Feb;15(2):175-84. doi: 10.1111/dom.12032. Epub 2012 Dec 3. PMID 23130654
- [Result] Gough SC, Bhargava A, Jain R, Mersebach H, Rasmussen S, Bergenstal RM. Low-volume insulin degludec 200 units/ml once daily improves glycemic control similarly to insulin glargine with a low risk of hypoglycemia in insulin-naive patients with type 2 diabetes: a 26-week, randomized, controlled, multinational, treat-to-target trial: the BEGIN LOW VOLUME trial. Diabetes Care. 2013 Sep;36(9):2536-42. doi: 10.2337/dc12-2329. Epub 2013 May 28. PMID 23715753
- [Result] Heller S, Mathieu C, Kapur R, Wolden ML, Zinman B. A meta-analysis of rate ratios for nocturnal confirmed hypoglycaemia with insulin degludec vs. insulin glargine using different definitions for hypoglycaemia. Diabet Med. 2016 Apr;33(4):478-87. doi: 10.1111/dme.13002. Epub 2015 Dec 13. PMID 26484727
- [Result] Vora J, Christensen T, Rana A, Bain SC. Insulin degludec versus insulin glargine in type 1 and type 2 diabetes mellitus: a meta-analysis of endpoints in phase 3a trials. Diabetes Ther. 2014 Dec;5(2):435-46. doi: 10.1007/s13300-014-0076-9. Epub 2014 Aug 1. PMID 25081590
- [Result] Aye MM, Atkin SL. Patient safety and minimizing risk with insulin administration - role of insulin degludec. Drug Healthc Patient Saf. 2014 Apr 30;6:55-67. doi: 10.2147/DHPS.S59566. eCollection 2014. PMID 24812526
- [Result] Sorli C, Warren M, Oyer D, Mersebach H, Johansen T, Gough SC. Elderly patients with diabetes experience a lower rate of nocturnal hypoglycaemia with insulin degludec than with insulin glargine: a meta-analysis of phase IIIa trials. Drugs Aging. 2013 Dec;30(12):1009-18. doi: 10.1007/s40266-013-0128-2. PMID 24170235
- [Result] Einhorn D, Handelsman Y, Bode BW, Endahl LA, Mersebach H, King AB. PATIENTS ACHIEVING GOOD GLYCEMIC CONTROL (HBA1c <7%) EXPERIENCE A LOWER RATE OF HYPOGLYCEMIA WITH INSULIN DEGLUDEC THAN WITH INSULIN GLARGINE: A META-ANALYSIS OF PHASE 3A TRIALS. Endocr Pract. 2015 Aug;21(8):917-26. doi: 10.4158/EP14523.OR. Epub 2015 Jun 29. PMID 26121451
- [Result] Russell-Jones D, Gall MA, Niemeyer M, Diamant M, Del Prato S. Insulin degludec results in lower rates of nocturnal hypoglycaemia and fasting plasma glucose vs. insulin glargine: A meta-analysis of seven clinical trials. Nutr Metab Cardiovasc Dis. 2015 Oct;25(10):898-905. doi: 10.1016/j.numecd.2015.06.005. Epub 2015 Jun 18. PMID 26232910
- [Result] Vora J, Seufert J, Solberg H, Kinduryte O, Johansen T, Hollander P. Insulin degludec does not increase antibody formation versus insulin glargine: an evaluation of phase IIIa trials. Diabetes Obes Metab. 2016 Jul;18(7):716-20. doi: 10.1111/dom.12621. Epub 2016 Feb 8. PMID 26663320
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 106 sites in 8 countries: Canada (11), France (6), Ireland (3), Russian Federation (7), South Africa (4), Ukraine (2), United Kingdom (18) and United States of America (55).
Pre-assignment Details: Subjects continued on metformin with or without dipeptidyl peptidase-4 (DPP-4) inhibitors at the pre-randomisation dose level and dosing frequency.
Groups:
- IDeg 200 U/mL OD: Insulin degludec (IDeg) 200U/mL was given once daily (OD) subcutaneously with the main evening meal in combination with metformin with or without dipeptidyl peptidase-4 (DPP-4) inhibitor treatment for 26 weeks.
- IGlar OD: Insulin glargine (IGlar) was given once daily (OD) subcutaneously according to approved labelling in combination with metformin with or without dipeptidyl peptidase-4 (DPP-4) inhibitor treatment for 26 weeks.
Period: Overall Study
Arm/Group | IDeg 200 U/mL OD | IGlar OD
Started | 230 | 230
Full Analysis Set | 228 (Two subjects were withdrawn because the subjects were randomised in error.) | 229 (One subject was withdrawn because the subject was randomised in error.)
Exposed | 228 | 228 (One subject withdrew prior to exposure to trial drug.)
Completed | 200 | 201
Not Completed | 30 | 29
Not completed — Adverse Event | 5 | 4
Not completed — Lack of Efficacy | 0 | 2
Not completed — Protocol Violation | 5 | 2
Not completed — Withdrawal Criteria | 3 | 9
Not completed — Other | 17 | 12

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all randomised subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg 200 U/mL OD | IGlar OD | Total
Number analyzed (Participants) | 228 | 229 | 457
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (9.0) | 57.3 (9.4) | 57.5 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 105 | 214
  Male | 119 | 124 | 243
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.3 (1.0) | 8.2 (0.9) | 8.3 (0.9)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 9.6 (2.9) | 9.7 (2.6) | 9.6 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline in HbA1c after 26 weeks of treatment
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects and missing data was imputed using last observation carried forward (LOCF). 2 subjects were withdrawn prior to exposure to the study drug in the IDeg arm as they were randomised in error and 1 subject in the IGlar arm.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg 200 U/mL OD | IGlar OD
Number analyzed (Participants) | 228 | 229
percentage of glycosylated haemoglobin | -1.30 (1.04) | -1.32 (0.98)

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change from baseline in FPG after 26 weeks of treatment
Time Frame: Week 0, Week 26
Population: The FAS included all randomised subjects and missing data was imputed using last observation carried forward (LOCF). For 3 subjects baseline values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg 200 U/mL OD | IGlar OD
Number analyzed (Participants) | 228 | 226
mmol/L | -3.70 (3.06) | -3.38 (2.96)

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 26 weeks + 7 days follow up
Description: Safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDeg 200 U/mL OD | IGlar OD
Serious Adverse Events (participants affected / at risk) | 15/228 | 10/228
Other Adverse Events (participants affected / at risk) | 51/228 | 60/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg 200 U/mL OD (N=228) | IGlar OD (N=228)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 4 (4) | 0 (0)
Polyp (General disorders) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic shock (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg 200 U/mL OD (N=228) | IGlar OD (N=228)
Diarrhoea (Gastrointestinal disorders) | 17 (24) | 19 (22)
Nasopharyngitis (Infections and infestations) | 17 (18) | 12 (13)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 15 (18)
Headache (Nervous system disorders) | 20 (27) | 24 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.